CLINICAL TRIAL: NCT05518019
Title: An Exploratory Investigation of a CBD Supplement's Impact on Sleep, Stress, and Focus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prima CBD (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20236
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Fear; Stress; Low Mood; Sleep
Keywords: Anxiety; Fear; Stress; Low Mood; Sleep; Focus; Calmness
MeSH Terms: conditions — Anxiety Disorders; Consciousness Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prima CBD "The Daily" Supplement (Experimental): Participants are provided with the dietary supplement (1 capsule per day). Participants are to take the supplement at the same time every day Participants will take a weekly well-being survey Participants are to complete the well-being questionnaire after the 4th week
  Interventions: Dietary Supplement: The Daily Supplement

INTERVENTIONS:
Dietary Supplement: The Daily Supplement — Each serving of the dietary supplement (defined as 1 softgel) contains the following formulation:
  Organic Broad Spectrum Hemp Extract 35mg Bio-Terpene Complex 52mg Palm Monoglycerides Organic Hemp Seed Oil, Clove Bud Oil, Black Pepper Berry Essential Oil Curcumin (Turmeric Root) Essential Oil
  Inactive ingredients: Organic Flaxseed Oil, Gel Shell (Modified Tapioca Starch, Glycerin, Purified Water, Maltitol

SUMMARY:
A high-quality broad-spectrum cannabidiol supplement with a bio-terpene complex will be administered once daily. It is hypothesized that this supplement will lead to improvements in sleep, focus, and stress. Previous research supports that CBD supplementation provides support to the endocannabinoid system, allowing the brain to better control negative psychological outcomes like fear, stress, and negative mood states.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Ability to take oral medication and be willing to adhere to the dietary supplement regimen (1 capsules per day).
* Must be in general good health (e.g., no long term health issues that would impact your participation.
* Moderate self-reported issues with stress, mood, focus, and sleep.

Exclusion Criteria:

* Current use of selective serotonin reuptake inhibitors or prescription medication for the treatment of depression or anxiety and have not been on a stable dose for more than 60 days.
* Currently receiving other psychotherapeutic treatment for anxiety or depression.
* Diagnosed anxiety or depression
* BMI over 40
* Known allergic reactions that would require the use of an epi-pen
* Females who are pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change in stress and anxiety as measured by questionnaires. | 2 months
  Feeling states that will be measured include stress, calmness, balance, relaxation, and focus
  Each endpoint will be reported by the participant on a 7-point scale of perceived frequency and severity of feeling states (Ranging from "Never" to "Everyday", and "None" to "Very severe")
Change in mood as measured by questionnaire | 2 months
  Feeling states that will be measured include stress, calmness, balance, relaxation, and focus
  Each endpoint will be reported by the participant on a 7-point scale of perceived frequency and severity of feeling states (Ranging from "Never" to "Everyday", and "None" to "Very severe")

SECONDARY OUTCOMES:
Change in sleep quality and quantity as measured by digital wearable devices and by self-report | 2 months
  Sleep will be measured two ways. Questionnaires will be used to assess sleep quality and quantity.
  Participants will also use wearable devices to track their sleep over the course of the study.

OTHER OUTCOMES:
Change in overall well-being as measured by self-report and questionnaires. | 2 months
  Each endpoint will be reported by the participant on a 7-point scale of perceived frequency and severity of feeling states (Ranging from "Never" to "Everyday", and "None" to "Very severe")

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided